CLINICAL TRIAL: NCT03159624
Title: Use of Porcine Small Intestinal Submucosa (SIS) Graft to Aid in Nasal Septal Remucosalization and Tissue Healing in Patients Following Use of Nasoseptal Flap Elevation for Skull Base Surgery
Brief Title: Nasal Septal Flap for Donor Site Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Stanford University (Other); Cook Group Incorporated (Industry)
Responsible Party: Principal Investigator, Brad Woodworth, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F140612003
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Results first posted 2019-09-16 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2019-08

CONDITIONS: Nasal Septum Perforation
Keywords: nasoseptal flap; tissue repair; wound healing; remucosalization; upper airway; granulation tissue; tissue graft
MeSH Terms: conditions — Nasal Septal Perforation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): 2x3 cm Biodesign™ SIS graft placement + overlying Doyle silastic sheet placement over the resulting exposed septum cartilage/bone
  Interventions: Other: Biodesign™ SIS graft; Other: Doyle silastic sheet
- Control Group (Active Comparator): Thin Doyle silastic sheet placement alone over the resulting exposed septum cartilage/bone
  Interventions: Other: Doyle silastic sheet

INTERVENTIONS:
Other: Biodesign™ SIS graft — 2x3 cm Biodesign™ SIS perforated mesentery graft
  Arms: Treatment Group
Other: Doyle silastic sheet — Doyle silastic sheet

SUMMARY:
The purpose of this study is to demonstrate the utility of porcine small intestinal submucosa (SIS) as a graft material that may aid in the natural healing process of freshly exposed bone and cartilage in the nasal cavity.

DETAILED DESCRIPTION:
Patients who undergo endoscopic endonasal skull base surgery, and may require nasoseptal flap placement as part of skull base reconstruction, will be informed, consented and enrolled for participation. If the intraoperative decision is ultimately made for harvest and placement of full-length nasoseptal flap by each individual surgeon, patients will then be consecutively, sequentially randomized to use of either:

* Thin Doyle silastic sheet placement alone over the resulting exposed septum cartilage/bone (20 randomly assigned patients)
* 2x3 cm Biodesign™ SIS perforated mesentery graft surface placement plus overlying Doyle silastic sheet placement over the resulting exposed septum cartilage/bone. (20 randomly assigned patients)

When used, Biodesign graft will be soaked in sterile saline out of the packaging, and placed as an intact single sheet over the exposed bone nasal septum bone/cartilage (without trimming). For uniformity and ease of future analysis, the bottom edge of the graft will be placed parallel to, and proximal to, the nasal floor cut edge remnant mucosal surface as possible. Except for a thin Doyle silastic sheet to cover the graft site, no additional reinforcement (suture/tissue glue) will be placed for those patients in the Biodesign graft arm.

Time Points and Study Parameters:

* All enrolled patients will have Doyle silastic sheeting removed only at 2 weeks post-op.
* All patients will receive 250cc normal saline topical nasal rinses starting at 14 days until 120 days post-op.
* No topical irrigation additives (budesonide/mupirocin) will be administered over 12 weeks.

All patients will be assessed at 2 weeks, 6 weeks and 12 weeks following randomization and entry into this study.

ELIGIBILITY:
Inclusion Criteria:

* Elective transnasal endoscopic skull base surgery where closure with a large nasoseptal flap (NSF) is anticipated (exposure of >75% of the ipsilateral nasal septum bone/cartilage)
* Patients without nutritional compromise or otherwise debilitated
* Patients who are able to consent for themselves

Exclusion Criteria:

* Bilateral nasoseptal flap (NSF) placement in the same operative setting
* Patients without significant bone/cartilage exposure to incorporate an intact 2x3 cm graft
* Patients requiring 24 hour supplemental oxygen via nasal cannula
* Patients who cannot consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Woodworth, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nayak JV, Rathor A, Grayson JW, Bravo DT, Velasquez N, Noel J, Beswick DM, Riley KO, Patel ZM, Cho DY, Dodd RL, Thamboo A, Choby GW, Walgama E, Harsh GR, Hwang PH, Clemons L, Lowman D, Richman JS, Woodworth BA. Porcine small intestine submucosal grafts improve remucosalization and progenitor cell recruitment to sites of upper airway tissue remodeling. Int Forum Allergy Rhinol. 2018 Oct;8(10):1162-1168. doi: 10.1002/alr.22156. Epub 2018 Jun 1. PMID 29856526

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 21 | 26
Completed | 21 | 25
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 21 | 26 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 23 | 39
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 6 | 11 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Post-operative Remucosalization at the Donor Site
Description: Mean change as measured by Visual Analogue Scale (VAS) scores from 3 independent reviewers from endoscopy videos collected at 2, 6, and 12 weeks. The Visual Analogue Scale for mean change in post-operative remucosalization is a Likert scale ranging from 0% (no remucosalization) to 100% (complete remucosalization), with higher scores representing better healing.
Time Frame: 2 weeks, 6 weeks, 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of remucosalization
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 21 | 26
percentage of remucosalization
  2 weeks | 47.8 [40.3 to 55.3] | 37.8 [31.1 to 44.5]
  6 weeks | 49.7 [41.6 to 57.8] | 43.5 [36.7 to 50.3]
  12 weeks | 73.9 [63.8 to 83.9] | 65.3 [56.97 to 73.7]
  overall change | 57.1 [52.1 to 62.2] | 48.9 [45.1 to 52.7]

2. Primary Outcome: Mean Change in Post-operative Locoregional Crusting at Donor Site
Description: Mean change as measured by Visual Analogue Scale (VAS) scores from 3 independent reviewers from endoscopy videos collected at 2, 6, and 12 weeks. The Visual Analogue Scale for mean change in post-operative crusting is a Likert scale ranging from 0 (no crusting) to 10 (complete crusting), with lower scores representing better healing.
Time Frame: 2 weeks, 6 weeks, 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 21 | 26
score on a scale
  2 weeks | 3.50 [2.99 to 4.01] | 4.22 [3.50 to 4.94]
  6 weeks | 4.22 [3.03 to 5.41] | 5.2 [4.17 to 6.24]
  12 weeks | 2.64 [1.48 to 3.80] | 2.92 [2.17 to 3.66]
  overall change | 3.45 [2.97 to 3.93] | 4.11 [3.63 to 4.59]

3. Primary Outcome: Mean Change in Post-operative Edema at the Donor Site
Description: Mean change as measured by Visual Analogue Scale (VAS) scores from 3 independent reviewers from endoscopy videos collected at 2, 6, and 12 weeks. The Visual Analogue Scale for mean change in post-operative edema is a Likert scale ranging from 0 (no edema) to 10 (severe edema), with lower scores representing better healing.
Time Frame: 2 weeks, 6 weeks, 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 21 | 26
score on a scale
  2 weeks | 3.34 [2.94 to 3.75] | 3.52 [3.16 to 3.89]
  6 weeks | 3.25 [2.74 to 3.76] | 3.15 [2.75 to 3.55]
  12 weeks | 2.26 [1.84 to 2.70] | 2.65 [2.11 to 3.19]
  overall change | 2.95 [2.73 to 3.18] | 3.11 [2.86 to 3.35]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/26
Other Adverse Events (participants affected / at risk) | 7/21 | 8/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=21) | Control Group (N=26)
minor septal perforation (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
development of transverse synechiae between septum and inferior turbinate (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No